CLINICAL TRIAL: NCT06364488
Title: TrueBlue Clinical Study - Investigating the Use of a Mobile Phone App TrueBlue for Monitoring Depression and Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BlueSkeye AI (Industry)
Collaborators: Institute of Mental Health Nottingham (Other); Nottinghamshire Healthcare NHS Trust (Other Government); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 295721
Record Dates: First submitted 2024-03-21; First posted 2024-04-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Depression; Depression, Postpartum; Anxiety in Pregnancy; Anxiety; Anhedonia; Perinatal Depression
Keywords: Depression; Anxiety; Perinatal
MeSH Terms: conditions — Depression; Depression, Postpartum; Anxiety Disorders; Anhedonia

STUDY DESIGN:
Intervention Model Description: 125 participants, of whom 12 will enter the initial 5-month within-study pilot phase aimed at understanding any device-related adverse events and usability issues.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Related Adverse Events (Other): The primary aim of the study is to demonstrate that use of the TrueBlue app to monitor depression is safe
  Interventions: Device: TrueBlue App

INTERVENTIONS:
Device: TrueBlue App — The use of the TrueBlue App, to generate automated measures of mood that can be assessed for agreement with validated clinical scales eg. PHQ9.

SUMMARY:
This trial will assess the safety, feasibility, acceptability, usability and agreement with validated scales of an automated mood monitoring App (TrueBlue), in adult, perinatal participants (recruited between 12 weeks of pregnancy and 12 weeks post-partum), recruited across multiple sites in Nottinghamshire, United Kingdom (UK). An initial within-study pilot phase will assess key aspects of the study including recruitment rate, usability issues and a detailed understanding of any device related adverse events; prior to full recruitment of a total 125 participants over a total 14-month period.

DETAILED DESCRIPTION:
This early-phase study of the TrueBlue App will recruit participants from Nottinghamshire Healthcare NHS Foundation Trust (NHFT), Nottingham University Hospitals NHS Trust (NUH) and a number of Primary Care sites in Nottinghamshire, UK. At study inclusion participants will be at least 18 years old, in the perinatal phase (between 12 weeks of pregnancy and 12 weeks post-partum), able to give capacious consent and satisfying the other detailed inclusion/exclusion criteria provided below. Initial recruitment will be to a 5-month, within-study pilot phase during which up to 12 participants will use the TrueBlue App for a 12-week period. Participants will be asked to complete two tasks on the App each week, involving reading or speaking to the App whilst it records the user's face and voice; and to complete each of the following four validated scales every two weeks: Patient Health Questionnaire 9-item scale (PHQ9), Edinburgh Postnatal Depression Scale (EPDS), Generalized Anxiety Disorder 7-item scale (GAD7), Temporal Experience of Pleasure Scale (TEPS). Adverse Events (AEs) will be detected through structured surveillance at weeks 6 and 12, in addition to encouraging participants to report any new or recurrent health problems during their period of App use. AEs will be assessed for plausibility of relatedness to App use [Device-Related Adverse Events; (DRAEs)], seriousness and expectedness; with discussion at the Trial Management Committee (TMC) focusing on developing any necessary mitigations, including technological or informational changes. The Standard Operating Procedure (SOP) for investigation of AEs includes a break to recruitment if serious DRAEs are identified. During the 5-month within-study pilot phase, stakeholder focus groups will be convened, separately for clinicians and patients, with up to 6 participants in each group focusing on AEs, usability issues, integration into care, liaison with Perinatal Psychiatry services and study governance. These sessions will be conducted by the study team, with recorded, anonymised transcripts subjected to thematic or content analysis depending on the depth of data. Anonymised reports from these focus groups will inform the TMC and the later individual, semi-structured interviews.

Following the 5-month within-study pilot phase and any necessary adjustments to SOPs (notified appropriately to the REC), we will enter a 9-month study period to full recruitment (125 participants). In this later period, as in the pilot phase, participants will use the TrueBlue App for up to 12 weeks, as described above, with continued surveillance for AEs including the 6 and 12 week reviews. Throughout the total 14-month study metrics will be collected on usability, feasibility and acceptability, alongside the validated self-completion questionnaires assessing depression (PHQ9, EPDRS), anxiety (GAD-7) and anhedonia (TEPS). Audio-visual data recorded through the weekly tasks will be used to generate automated mood scores that will then be assessed for agreement with the validated scales.

Up to 30 study participants will also be invited to take part in individual, semi-structured interviews assessing their experience of the app, including barriers and facilitators to use. Recruitment will be to saturation of themes, or to a maximum of 30 interviews, using purposive sampling to encourage a representation of participants with high and low System Usability Scale (SUS) scores. Interview transcripts will be subjected to thematic analysis.

This study has received approval from the relevant UK ethics committee (NHS Rec reference 22/LO/0009, IRAS project reference: 295721) and regulatory authority (MHRA, CI/2023/0063/GB).

ELIGIBILITY:
Inclusion Criteria:

- 18 years or older

* Fluent in spoken and written English
* Has capacity to provide consent
* At least 12 weeks pregnant or less than 12 weeks postpartum
* Access to internet connectivity
* Access to a compatible smart phone device (for up to 10 participants, where needed through not having a personal device, this access may be provided through the study team).
* Has a current GP within Nottinghamshire

Exclusion Criteria:

* ● Current clinically diagnosed psychiatric disorder other than depression

  * Previous history of a clinically diagnosed psychiatric disorder, other than depression and generalised anxiety disorder (including previous Psychosis, Bipolar Disorder, Personality Disorder, Substance Abuse Disorders, Eating Disorders)
  * Clinical diagnosis of an Autistic Spectrum Disorder, Attention Deficit Hyperactivity Disorder, Parkinson's Disease or other current Neurological Disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of device related adverse events | up to12 weeks
  Percentage of participants who experience at least one device related adverse event during the 12-week period from baseline to end of app use (ascertained through both voluntary reporting and active surveillance at 6 and 12 weeks).

SECONDARY OUTCOMES:
Rate of initial use (assessing feasibility and acceptability) | up to12 weeks
  Rate of initial community use (defined as at least one completed use after initial demonstration)
Rate of New Depression or Risk (Suicidality) events | up to12 weeks
  Percentage of participants who generate amber or red flag warnings through inputs to validated depression measures (PHQ9, EPDRS)
Rate of referral to Perinatal Psychiatry services | up to12 weeks
  Percentage of patients referred to Perinatal Psychiatry services, based on study team assessment of amber or red flag warnings.
Rate of acceptance of referrals to Perinatal Psychiatry | up to12 weeks
  Rate of referred patients who are subsequently accepted by Perinatal Psychiatry services.
Diagnosis rate for depression, or other mental health problems, during the period of study. | 14 months
  Rate of patients diagnosed with a new or recurrent episode of depression, or other mental health problem during the period of study. Rate of these events picked up through App use (and Perinatal Psychiatry referral system).
Continued use (acceptability) | up to12 weeks
  Frequency of device usage by participants, following initial use in the community
Loss to follow-up | 14 months
  Rate of loss to follow-up within study.
Usability (quantitative measure) | up to12 weeks
  Analysis of System Usability Scale (SUS) score at following completion of app use (minimum value= 0, maximum value = 100).
Agreement between TrueBlue generated score and validated scales | 14 months
  Assessment of the agreement between TrueBlue generated scores (through processed audio-visual data) and the validated scales (PHQ9, EPDS, GAD7, TEPS).
Thematic results | 14 months
  Results from thematic analyses of transcripts from stakeholder meetings and individual semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Nixon, MBBS, Principal Investigator — School of Medicine, University of Nottingham and Nottinghamshire Healthcare NHS Trust
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No
To comply with the data protection act, personal data will be deleted as soon as possible after it is no longer needed for the study.

REFERENCES:
- [Background] Braun V, Clarke V. Toward good practice in thematic analysis: Avoiding common problems and be(com)ing a knowing researcher. Int J Transgend Health. 2022 Oct 25;24(1):1-6. doi: 10.1080/26895269.2022.2129597. eCollection 2023. No abstract available. PMID 36713144
- [Background] Gard D, Gard M, Kring A, John O. Anticipatory and consummatory components of the experience of pleasure: A scale development study. J Res Pers. 2006;40:1086-110
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qualitative research in psychology. 2006 Jan 1;3(2):77-101.
- [Background] Brooke J. SUS-A quick and dirty usability scale. Usability evaluation in industry. 1996 Jun 11;189(194):4-7.